CLINICAL TRIAL: NCT06116409
Title: Efficacy of Modified Thoracoabdominal Nerves Block Through Perichondrial Approach in Total Laparoscopic Hysterectomies on Postoperative Pain
Brief Title: Efficacy of Modified Thoracoabdominal Nerves Block Through Perichondrial Approach in Total Laparoscopic Hysterectomies
Status: Completed | Type: Observational
Sponsor: Dr. Lutfi Kirdar Kartal Training and Research Hospital (Other Government)
Responsible Party: Principal Investigator, kübra taşkın, specialist medical doktor, Dr. Lutfi Kirdar Kartal Training and Research Hospital
Other Study IDs: DrLutfiKirdarANESTHESİA
Record Dates: First submitted 2023-10-20; First posted 2023-11-03 (Actual); Last update posted 2025-02-25 (Actual); Status verified 2025-02

CONDITIONS: Postoperative Pain
MeSH Terms: conditions — Pain, Postoperative | interventions — Bupivacaine

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- M-TAPA GROUP: Group 1 patients will receive a modified thoracoabdominal nerve block (M-TAPA) with a perichondrial approach using 40 ml of 0.25% bupivacaine guided by ultrasound (US).
  Interventions: Drug: Bupivacain
- CONTROL GROUP: Patients in Group 2 (the control group) will receive routine multimodal analgesia, which includes tramadol at a dose of 1 mg/kg and paracetamol at a dose of 15 mg/kg.

INTERVENTIONS:
Drug: Bupivacain — Bupivacaine was used for postoperative analgesia block.
  Groups: M-TAPA GROUP

SUMMARY:
TAPA is a new analgesic block technique that involves the injection of local anesthetics into the thoracoabdominal nerves using a perichondrial approach. Application to the undersurface of the rib cartilage is considered as Modified TAPA (M-TAPA). These techniques are commonly applied for postoperative analgesia in surgeries and are effective and safe when performed under ultrasound guidance.

DETAILED DESCRIPTION:
Between September 2023 and October 2023, a study will be conducted involving 50 elective total laparoscopic hysterectomy patients aged 18-65 with ASA (American Society of Anesthesiologists) physical status classification of 1-3. Patients with ASA status 4 or higher, aged 65 and above, under 18 years of age, those who have previously undergone laparotomy, or those with a known local anesthesia allergy will not be included in the study. Patients who require intubation and are admitted to the intensive care unit, or those who experience mortality, will be excluded from the study.

One day before surgery, all patients will undergo a preoperative assessment and provide written informed consent to participate in the study. Patients will be randomly assigned to groups using a computer-generated random table. In Group 1, patients will receive a modified thoracoabdominal nerve block (M-TAPA) with a perichondrial approach using 40 ml of 0.25% bupivacaine guided by ultrasound (US). In Group 2 (the control group), routine multimodal analgesia (tramadol 1 mg/kg, paracetamol 15 mg/kg) will be administered. The needle-like spread of bupivacaine or saline beneath the undersurface of the rib cartilage, observed under US, will indicate the success of the procedure. These procedures will be performed postoperatively. At the end of the surgery, both groups will receive 1 mg/kg tramadol IV and 15 mg/kg paracetamol IV for analgesia.

Demographic data, medical history, ASA classification, and the presence of coronary artery disease (CAD) and overactive bladder (OAB) before and after M-TAPA, anesthesia time, surgical duration, time to tracheal extubation (time after skin closure), total remifentanil and muscle relaxant doses, total fluid administered, urine volume, and the total volume of allogeneic erythrocytes and plasma infused during the surgery will be recorded. Additionally, postoperative hypotension development (systolic blood pressure dropped more than 30% from baseline or SBP < 80 mmHg before anesthesia), nausea and vomiting, hypoxemia (SpO2 < 90% or PaO2 < 60 mmHg), hypercapnia (PaCO2 > 45 mmHg), and agitation during the waking period will be recorded.

In the ward, 2*1 non-steroidal anti-inflammatory drugs (NSAIDs) will be administered for analgesia. Numerical Rating Scale (NRS) will be assessed postoperatively at 2, 6, 12, and 24 hours, and tramadol consumption will be recorded. A numerical rating scale (NRS) ranging from 0 (no pain) to 10 (worst imaginable pain) will be used for pain assessment. If NRS is greater than 4, rescue analgesia with tramadol will be administered. After surgery, all patients will be transferred to the post-anesthesia care unit (PACU).

ELIGIBILITY:
Inclusion Criteria:

* electively total laparoscopic hysterectomy operations

  * ASA II-III,
  * between 18-65 years

Exclusion Criteria:

* ASA IV and above • over 65 - under 18 years of age allergy to local anesthetics

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Between September and November 2023, 50 patients aged 18-65 with ASA (American Society of Anesthesiologists) physical status classification of I-III, who are scheduled to undergo elective total laparoscopic hysterectomy, will participate in the study.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2023-09-01 (Actual); Primary Completion 2023-11-24 (Actual); Study Completion 2023-11-30 (Actual)

PRIMARY OUTCOMES:
Evaluate patients' postoperative pain | postoperative 24 hours
  The primary aim of this study is to evaluate and compare the postoperative analgesic effectiveness of modified thoracoabdominal nerve block (M-TAPA) in total laparoscopic hysterectomy. Numerical rating scale (NRS) will be used for postoperative analgesic effectiveness. NRS ranging from 0 (no pain) to 10 (worst imaginable pain) will be used for pain assessment. If NRS is greater than 4, rescue analgesia with tramadol will be administered.

CONTACTS AND LOCATIONS:
Overall Officials: hülya yılmaz ak, Principal Investigator — Kartal Dr Lutfi Kırdar City Hospital
Locations (1):
- University of Health Science, Kartal Dr Lütfi Kırdar Training and Research Hospital, Istanbul, İ̇stanbul, Turkey (Türkiye)